CLINICAL TRIAL: NCT01297192
Title: An Open-label, One-sequence, Two-arm Study to Evaluate the Effect of Steady State Concentrations of Mirabegron on the Pharmacokinetics of Solifenacin and to Evaluate the Effect of Steady State Concentrations of Solifenacin on the Pharmacokinetics of Mirabegron in Healthy Young Male and Female Subjects
Brief Title: A Clinical Study to Assess the Effect on Pharmacokinetics of Dosing Mirabegron (YM178) and Solifenacin Simultaneously
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 178-CL-069; 2008-007929-40 (EudraCT Number)
Record Dates: First submitted 2011-02-15; First posted 2011-02-16 (Estimated); Last update posted 2013-07-29 (Estimated); Status verified 2013-07

CONDITIONS: Healthy Volunteers; Pharmacokinetics of Mirabegron
Keywords: YM178; Mirabegron; DDI; Phase I; Solifenacin; Pharmacokinetics; Pharmacokinetics of mirabegron
MeSH Terms: interventions — Solifenacin Succinate; mirabegron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Arm 1 (Other): The effect of mirabegron on the pharmacokinetics of solifenacin
  Interventions: Drug: solifenacin succinate; Drug: mirabegron
- Treatment Arm 2 (Other): The effect of solifenacin on the pharmacokinetics of mirabegron
  Interventions: Drug: solifenacin succinate; Drug: mirabegron

INTERVENTIONS:
Drug: solifenacin succinate — Oral
  Other Names: Vesicare; YM905
Drug: mirabegron — Oral
  Other Names: YM178

SUMMARY:
This study investigates whether mirabegron (YM178) has an effect on the pharmacokinetics of solifenacin and whether solifenacin has an effect on the pharmacokinetics of mirabegron.

ELIGIBILITY:
Inclusion Criteria:

* Male subject must agree to sexual abstinence and/or use a highly effective method of birth control from screening until 3 months after last dose of study medication
* Female subject must be of non-child bearing potential, i.e. post menopausal, surgically sterilized (e.g. tubal ligation), hysterectomy in medical history, or must practice an adequate non-hormonal contraceptive method to prevent pregnancies. Non-hormonal contraceptive methods are defined as:

  * sexual abstinence from 1 month before admission until 3 months after discharge
  * subject's sexual partner has been surgically sterilized (since at least 3 months prior to the screening), or
  * subject is under two (2) of the following contraceptive methods: I. diaphragm with spermicide II. intrauterine device III. sexual partner is using condoms in combination with a spermicidal cream
* Body Mass Index between 18.5 and 30.0 kg/m2, inclusive

Exclusion Criteria:

* Known or suspected hypersensitivity to mirabegron or any of the components of the formulation used
* Known or suspected hypersensitivity to solifenacin succinate or any of the components of the formulation used
* Pregnant or breast feeding within 6 months before screening assessment.
* Any of the liver function tests (i.e. ALT, AST and Alkaline phosphatase) above the upper limit of normal at repeated measures
* Any clinical significant history of or at risk for urinary retention, severe gastro-intestinal condition (including toxic megacolon), myasthenia gravis or narrow-angle glaucoma
* Any clinically significant history of asthma, eczema, any other clinically significant allergic condition or previous severe hypersensitivity to any drug (excluding non-active hay fever)
* Any clinically significant history of any other disease or disorder - gastrointestinal, cardiovascular, respiratory, renal, hepatic, neurological, dermatological, psychiatric or metabolic as judged by the medical investigator
* Any clinically significant abnormality following the investigator's review of the pre-study physical examination, ECG and clinical laboratory tests
* Abnormal pulse and/or blood pressure measurements at the pre-study visit as follows: pulse <40 or >90 bpm; mean systolic blood pressure >140 mmHg; mean diastolic blood pressure >90 mmHg (blood pressure measurements taken in triplicate after subject has been resting in supine position for 5 min; pulse will be measured automatically)
* A marked baseline prolongation of QT/QTc interval after repeated measurement of >450 ms, a history of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmias or torsades de pointes, structural heart disease, or a family history of Long QT syndrome (LQTS)
* Use of any prescribed or OTC (over-the counter) drugs (including vitamins, oral contraceptives or hormone replacement therapy, natural and herbal remedies, e.g. St. John's wort) in the 2 weeks prior to admission to the Clinical Unit, except for paracetamol (up to 3 g/day)
* Regular use of any inducer of liver metabolism (e.g. barbiturates, rifampin) in the 3 months prior to admission to the Clinical Unit
* Any use of drugs of abuse within 3 months prior to admission to the Clinical Unit
* History of smoking more than 10 cigarettes (or equivalent amount of tobacco) per day within 3 months prior to admission to the Clinical Unit
* History of drinking more than 21 units of alcohol per week (1 unit=270 cc of beer or 40 cc of spirits or 1 glass of wine) (>14 units of alcohol for female subjects) within 3 months prior to admission to the Clinical Unit
* Donation of blood or blood products within 3 months prior to admission to the Clinical Unit
* Positive serology test for HBsAg, anti HAV (IgM), anti-HCV or anti-HIV 1+2
* Subject who, in the opinion of the investigator, is not likely to complete the trial for any reason
* Participation in any clinical study within 3 months or participation in more than 3 clinical studies within 12 months, prior to the expected date of enrolment into the study, provided that the clinical study did not entail a biological compound with a long terminal half life
* Any clinical condition, which, in the opinion of the investigator, would not allow safe completion of the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2009-03; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Assessment of pharmacokinetics of solifenacin through analysis of blood samples | Days 1 - 9 and Days 23 - 39
Assessment of pharmacokinetics of mirabegron through analysis of blood samples | Time Frame: Days 1 - 6 and Days 16 - 21

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma Europe B.V.
Locations (1):
- Paris, France